CLINICAL TRIAL: NCT03635645
Title: Experimental and Clinical Studies of Retinal Stimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, James Weiland, Professor of Biomedical Engineering, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HUM00122699; R01EY022931-05 (NIH)
Record Dates: First submitted 2018-07-26; First posted 2018-08-17 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Retinal stimulation (Experimental): Alternative stimulus patterns will be tested (vs. baseline). The intervention is the alternative stimulus pattern. The intervention will be tested only in the clinic vs. baseline. The subject will go home with baseline settings. The two alternative stimulus patterns to be tested are asymmetric waveforms and bipolar stimulus.
  Interventions: Device: New visual processing unit (VPU) with asymmetric waveforms; Device: New VPU with bipolar stimulation

INTERVENTIONS:
Device: New visual processing unit (VPU) with asymmetric waveforms — A VPU will apply asymmetric and symmetric stimulation pulses.
Device: New VPU with bipolar stimulation — A VPU will apply bipolar stimulus pulses.

SUMMARY:
The study will evaluate new methods of retinal stimulation and training with the goal of improving the visual ability of retinal prosthesis participants.

DETAILED DESCRIPTION:
The study will test new ways to make the retinal prosthesis visual perception easier with auditory-visual training and how to make the retinal prosthesis work better at perceiving shapes.

ELIGIBILITY:
Inclusion Criteria:

* Must be implanted with an Argus II Retinal Prosthesis system.
* Have 5 or more electrodes that create a perception with stimulation.
* Must be willing and able to comply with the protocol testing requirements.

Exclusion Criteria:

* Subjects participating in another investigatory drug or device study
* Any disease or condition that prevents understanding or communication of informed consent, study demands, and testing protocols.

Ages: 25 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-10-30 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Percent change in stimulus thresholds | Baseline, 8 hours
  Compare baseline threshold with threshold of modified stimulus parameters. Threshold is measured in microCoulumbs ( the product of stimulus duration and stimulus amplitude).
Change in shape perception | Baseline, 8 hours
  As measured by elongation ratio. The elongation ratio is the ratio of major axis length to minor axis length of an ellipse. Subjects will draw shapes on a touch screen and these shapes will be fit to an ellipse.

CONTACTS AND LOCATIONS:
Overall Officials: James Weiland, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States